CLINICAL TRIAL: NCT05352308
Title: The Evaluation of a Narrative Communication Intervention to Increase Human Papillomavirus Vaccination Intentions and Uptake in a Hispanic-Majority College Population
Brief Title: Evaluation of a Narrative Communication Intervention to Increase Human Papillomavirus Vaccination Intentions and Uptake
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sara Fleszar (Other)
Responsible Party: Sponsor-Investigator, Sara Fleszar, Principal Investigator, University of California, Merced
Organization: University of California, Merced (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UCM2021-142
Record Dates: First submitted 2022-04-18; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Human Papilloma Virus; Intention; Behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Common Sense Model Guided Narrative Video Group (Experimental): The narrative videos is guided by the CSM and designed to provide a comprehensive resource for college students. The narrative video addresses illness risk representations and information on HPV, the HPV vaccine, and HPV-related cancers. The format of the narrative video includes (1) a direct testimonial of a college woman (in her dorm room) telling a story to her roommates about what motivated her to get vaccinated, and (2) a conversation among the roommates where information about the HPV vaccine is discussed.
  Interventions: Behavioral: Common Sense Model Guided Narrative Video
- Standard of Care Group (No Intervention): Participants in the standard of care group will receive the Centers for Disease Control and Prevention's Vaccine Information Statement (VIS; https://www.cdc.gov/vaccines/hcp/vis/vis-statements/hpv.pdf). The VIS contains information about HPV, the HPV vaccine, and the benefits and risks of the vaccine.
  The VIS will be utilized because healthcare providers are required to distribute the VIS to patients before receiving each dose of the HPV vaccine, it is easy to understand, and it is publicly available information.
- Time & Attention Group (No Intervention): Participants in the time and attention video group will receive a Centers for Disease Control and Prevention video on binge drinking (https://youtu.be/I9hdkDTaQWU; 4:22 minutes). The video contains information on the health risks of binge drinking including unintended pregnancy, sexually transmitted diseases, injury, car accidents, violence, and HIV/AIDS

INTERVENTIONS:
Behavioral: Common Sense Model Guided Narrative Video — The narrative video will address illness risk representations and information on HPV, the HPV vaccine, and HPV-related cancers
  Arms: Common Sense Model Guided Narrative Video Group

SUMMARY:
The current study aims to evaluate a newly developed CSM narrative intervention in increasing HPV vaccination intentions and uptake in adults aged 18 to 26 years. The efficacy of the newly designed CSM-guided narrative video will be compared against a time and attention video and the standard of care print educational materials in increasing the intentions and uptake of the HPV vaccine in an adult Hispanic-majority college population. It is expected that participants receiving the CSM-guided narrative video will have greater HPV vaccine intentions compared with participants in the time and attention video and standard of care print education material groups. It is also hypothesized that participants receiving the CSM-guided narrative video will have greater HPV vaccine uptake at one month post-intervention compared with participants in the time and attention video and standard of care print education material groups.

DETAILED DESCRIPTION:
The current study aims to evaluate a newly developed CSM narrative intervention in increasing HPV vaccination intentions and uptake in adults aged 18 to 26 years. The efficacy of the newly designed CSM-guided narrative video will be compared against a time and attention video and the standard of care print educational materials in increasing the intentions and uptake of the HPV vaccine in an adult Hispanic-majority college population.

Main Hypotheses:

H1. Participants receiving the CSM-guided narrative video will have greater HPV vaccine intentions compared with participants in the time and attention video and standard of care print education material groups.

H2. Participants receiving the CSM-guided narrative video will have greater HPV vaccine uptake at one month post-intervention compared with participants in the time and attention video and standard of care print education material groups.

Secondary Hypotheses:

H3: For participants receiving the CSM-guided narrative video compared with participants in the time and attention video and standard of care print education material, it is expected that there will be increases in illness risk perceptions, risk-action coherence, knowledge of the HPV and HPV vaccine, perceived effectiveness of the HPV vaccine, perceived severity and susceptibility of HPV and decreases in perceived harms of the HPV vaccine, barriers to the HPV vaccine, and uncertainty of the HPV vaccine immediately post-intervention as well as one month post-intervention.

H4. It is expected that the relationship between intervention groups (i.e., CSM-guided narrative video, time and attention video, standard of care print material) and vaccine uptake will be moderated by three sets of moderators: (1) knowledge of HPV and the HPV vaccine, illness risk perceptions, risk-action coherence, narrative engagement, and realism, (2) perceived effectiveness of the HPV vaccine, perceived severity and susceptibility of the HPV virus, and perceived harms of the vaccine, barriers to receiving the vaccine, and uncertainty of the vaccine, and (3) vaccine intentions.

H5. It is expected that permissive sexual behavior will moderate the relationship between the intervention groups (i.e., CSM-guided narrative video, time and attention video, standard of care print material) and vaccine intentions and uptake, and knowledge of HPV and the vaccine. Further, it is expected that this relationship will be moderated by religious commitment.

H6. It is expected that there will be a moderating effect of story-telling cultures (Hispanic/Latinx and/or African American/Black compared to non-Hispanic white participants) on the relationship between the intervention groups (i.e., CSM-guided narrative video, time and attention video, standard of care print material) and vaccine intentions and uptake, narrative engagement, and realism.

Participants will be recruited via the University's SONA system for course credits. Students aged 18-26 years who have not received any doses of the HPV vaccine are eligible to participate. After completing the study screener, eligible participants will be directed to Qualtrics, a web-based survey platform. Participants will be asked to provide informed consent and complete a baseline survey. Once the baseline survey is complete, participants will be contacted 2 days post-baseline survey completion. At two days post-baseline participants will be randomized via Qualtrics' Randomizer into either the CSM-guided narrative video, to a time and attention video (i.e., CDC video on binge drinking), or the standard of care print educational materials (i.e., Centers for Disease Control and Prevention's Vaccine Information Statement). Participants will then be directed to a post-intervention survey via Qualtrics. Participants in all groups will be asked to be contacted by the research team one-month post-intervention to assess if they received the HPV vaccine. If they have not received the HPV vaccine, their intentions to receive the vaccine will be assessed as well as the longer-term effects of the groups on illness risk representations, risk-action link coherence, knowledge of HPV and HPV vaccine, and effectiveness, harms, barriers, and uncertainty of the HPV vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate students enrolled in the university's SONA system
* Aged 18-26 years
* Have not received any doses of the HPV vaccine
* Have working audio (e.g., headphones/speakers)

Exclusion Criteria:

* Students who are not undergraduates
* Undergraduates not participating in the university's SONA system
* Aged <18 or >26 years
* Have received any dose/shot (1st, 2nd, or 3rd doses/shots) of the HPV vaccine
* Do not have working audio (e.g., headphones/speakers)

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-04-20 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to immediately post-intervention in intentions | Baseline to 2 days post-baseline
  Intentions will be assessed with a previous measure to assess behavioral intentions (α = .92 in a sample of young adults; Moyer-Guse, Chung, & Jain, 2011) which has been adapted for use to assess intentions to engage in several HPV-related behaviors (Landrau, 2020). The assessment asks participants, on a scale of 1 = definitely will not to 7 = definitely will, "What is the likelihood that you will": (1) "Get the HPV vaccine within the next 30 days" and (2) "Get the HPV vaccine within the next 12 months." Several other HPV-related behaviors are assessed by asking participants, "What is the likelihood that you will engage in the following behaviors over the next 6 months on a scale of 0 = definitely will not to 6 = definitely will." Sample statements include (1) "Discuss the HPV vaccine with a healthcare provider" and (2) "Search for more information about the HPV vaccine." Higher scores indicate higher intentions to engage in HPV-related behaviors.
Change from immediately post-intervention to one-month post-intervention in intentions | 2 days post-baseline to one month post-baseline
  Intentions will be assessed with a previous measure to assess behavioral intentions (α = .92 in a sample of young adults; Moyer-Guse, Chung, & Jain, 2011) which has been adapted for use to assess intentions to engage in several HPV-related behaviors (Landrau, 2020). The assessment asks participants, on a scale of 1 = definitely will not to 7 = definitely will, "What is the likelihood that you will": (1) "Get the HPV vaccine within the next 30 days" and (2) "Get the HPV vaccine within the next 12 months." Several other HPV-related behaviors are assessed by asking participants, "What is the likelihood that you will engage in the following behaviors over the next 6 months on a scale of 0 = definitely will not to 6 = definitely will." Sample statements include (1) "Discuss the HPV vaccine with a healthcare provider" and (2) "Search for more information about the HPV vaccine." Higher scores indicate higher intentions to engage in HPV-related behaviors.

SECONDARY OUTCOMES:
HPV Vaccine Uptake | one month post-baseline
  HPV vaccine uptake will be assessed at one and three months post-intervention. Participants will answer the follow-up question, "Have you received any dose of the HPV vaccine in the past one/three months? -that is, since the last time you completed a session for this study?". If a participant indicates that they have received a dose of the HPV vaccine, they will be asked, "What dose of the HPV vaccine have you completed"? Participants will respond by indicating 1 = 1st dose, 2 = 2nd dose, and 3 = 3rd dose. Participants will then be asked to identify the date (approximate date if exact date is unknown) that they received the dose(s) from a provided calendar. HPV vaccine uptake will be measured at 1-month post-intervention.
Change from baseline to immediately post-intervention in Knowledge of HPV and HPV Vaccine | baseline to 2 days post-baseline
  Participants' knowledge of HPV will be measured with 10 true/false statements adapted from Kester and colleague's (2014) HPV vaccine knowledge assessment developed for use in young adults. The measure is comprised of 5 true and 5 false statements. Participants can also indicate "I don't know" for each statement. A higher percentage correct indicates greater HPV and vaccine knowledge. Participants who identify a statement incorrectly will be considered "misinformed", and those who identify a statement with "I don't know" will be considered "uninformed" about that aspect of HPV or the vaccine.
Change from baseline to immediately post-intervention in Effectiveness, Harms, Barriers, & Uncertainty of HPV Vaccine | baseline to 2 days post-baseline
  The perceived effectiveness, harms, barriers, and uncertainty will be measured with an adapted version of the Carolina HPV Immunization Attitudes and Beliefs Scale (CHIAS). The CHIAS will be adapted for use with an adult population and targeted to information from the narrative video. The four subscales are (1) perceived potential harms from the vaccine; (2) perceived barriers to HPV vaccination including cost and access to a healthcare provider; (3) perceived effectiveness of the HPV vaccine against protecting against genital warts, cervical cancer, penial, anus, and head and neck cancers; and (4) uncertainty which includes not having enough information about the vaccine and perception of community vaccination norms. Participants will be asked to rate the agreement with the statement provided on a 7-point Likert scale with 0 = strongly disagree to 6 = strongly agree. Higher scores represent more agreement with the statements provided.
Change from baseline to immediately post-intervention in Perceived Severity & Susceptibility of the HPV Virus | baseline to 2 days post-baseline
  Perceived severity and susceptibility of the HPV virus will be measured with questions developed by Frank and Colleagues (2017). Perceived severity of the HPV virus will be measured with the question, "What impact do you think having the HPV infection would have on your life?" with responses on a scale ranging from 0 = no impact to 10 = severe impact. Perceived susceptibility of contracting the HPV virus will be measured with "What do you think your chances of getting the HPV infection are?" Responses were on a scale ranging from 0 = it will definitely not happen to me to 10 = this will definitely happen to me. Higher scores indicate higher perceived severity and susceptibility of contracting the HPV virus. Perceived severity and susceptibility of HPV will be measured at baseline and immediately post-intervention.
Change from baseline to immediately post-intervention in Illness Risk Representations | baseline to 2 days post-baseline
  The Assessment of Illness Risk Representations (AIRR; Cameron, 2008) will be used to measure the conceptual and concrete (imagery) HPV risk representations. The AIRR contains a subscale assessing imagery contents which have been adapted for use with assessing HPV virus risk representations. The AIRR also includes subscales that assess risk beliefs about identity, timeline, consequences, personal control, cause, and coherence which have been adapted from the revised illness perception questionnaire.
Change from immediately post-intervention to one-month post-intervention in Illness Risk Representations | 2 days post-baseline to one month post-baseline
  The Assessment of Illness Risk Representations (AIRR; Cameron, 2008) will be used to measure the conceptual and concrete (imagery) HPV risk representations. The AIRR contains a subscale assessing imagery contents which have been adapted for use with assessing HPV virus risk representations. The AIRR also includes subscales that assess risk beliefs about identity, timeline, consequences, personal control, cause, and coherence which have been adapted from the revised illness perception questionnaire.
Change from baseline to immediately post-intervention in Risk-Action Coherence | baseline to 2 days post-baseline
  Risk-action coherence or having a coherent understanding of the risk-action link between the risk of contracting HPV and receiving HPV vaccine will be assessed with a measure adapted from Bishop et al. (2005). Sample questions include, "I have a clear understanding of how the HPV vaccine can reduce the chance of contracting HPV" and "I would find it easy to explain to someone else how the HPV vaccine can protect from contracting HPV" with responses ranging from 0 = strongly disagree to 4 = strongly agree. Higher scores indicate a higher coherent understanding of the risk-action link between HPV risk and the HPV vaccine.
Change from immediately post-intervention to one-month post-intervention in Risk-Action Coherence | 2 days post-baseline to one month post-baseline
  Risk-action coherence or having a coherent understanding of the risk-action link between the risk of contracting HPV and receiving HPV vaccine will be assessed with a measure adapted from Bishop et al. (2005). Sample questions include, "I have a clear understanding of how the HPV vaccine can reduce the chance of contracting HPV" and "I would find it easy to explain to someone else how the HPV vaccine can protect from contracting HPV" with responses ranging from 0 = strongly disagree to 4 = strongly agree. Higher scores indicate a higher coherent understanding of the risk-action link between HPV risk and the HPV vaccine.
Narrative Engagement | 2 days post-baseline
  The narrative engagement will be measured with the 12-item Narrative Engagement Scale. This scale measures four interrelated subconstructs: (1) narrative understanding, or the comprehension of the narrative and ease of audience to construct meaning from the narrative (2) attentional focus which describes the non-conscious focus on the narrative; (3) emotional engagement, which measures the emotions that are evoked within the audience ; (4) narrative presence, which measures the loss of awareness of the self and the space produced by the narrative. Responses ranged from 1 = strongly disagree to 7 = strongly agree. Higher scores indicated higher engagement in the narrative. The narrative engagement scale was only assessed in the post-intervention survey.
Realism | 2 days post-baseline
  Realism was measured with 2-items, "The story in the video can happen in real life", and "The events in the video could have been inspired by real-life situations," which were adapted for use with adults from Soto-Sanfiel & Angulo-Brunet (2020). Both questions assess the plausibility of the narrative (i.e., the narrative could occur in real-life; Hall, 2003). Participants will be asked to what degree they agree with the statements above on a scale of 0= strongly disagree to 4= strongly agree, with higher scores indicating greater narrative realism.
Religious Commitment | baseline
  Religious commitment will be measured with the 10-item Religious Commitment Inventory-10 (RCI-10; Worthington et al., 2003). The RCI-10 assesses the level of religious commitment or the extent to which an individual adheres to their religious beliefs, values, and practices, using a 5-point Likert rating scale (1= not at all true of me to 5= totally true of me). Sample items include, "I spend time trying to grow in understanding of my faith." and "I enjoy spending time with others of my religious affiliation". Higher scores indicate greater religious commitment (α = 0.96; Birmingham et al., 2019).

CONTACTS AND LOCATIONS:
Overall Officials: Linda Cameron, PhD, Study Director — University of California, Merced

IPD SHARING:
Plan to Share IPD: Undecided